CLINICAL TRIAL: NCT01681017
Title: Global Network for Women's and Children's Health Research Does Implementation of HELPING BABIES BREATHE (HBB) Save Lives?
Brief Title: Global Network Implementation of Helping Babies Breathe (HBB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Laerdal Medical (Industry); Indiana University School of Medicine (Other); Christiana Care Health Services (Other); Massachusetts General Hospital (Other); Moi Univeristy (Other); Jawaharlal Nehru Medical College (Other); Lata Medical Research Foundation, Nagpur (Other); RTI International (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GN HBB Study
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Perinatal Mortality
Keywords: Perinatal Mortality; Asphyxia; Stillbirth; Neonatal Death; Resuscitation; Helping Babies Breathe; among births greater than one thousand five hundred grams
MeSH Terms: conditions — Perinatal Death; Asphyxia; Stillbirth | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Facilities (Other): Have appropriate staff trained in HBB and have HBB equipment provided
  Interventions: Other: HBB/ENC supplies
- Master Trainers (Other): Receive appropriate HBB training
  Interventions: Behavioral: HBB/ENC Training and Equipment
- Facilitators (Other): Receive appropriate HBB training
  Interventions: Behavioral: HBB/ENC Training and Equipment
- Learners (Other): Receive appropriate HBB training
  Interventions: Behavioral: HBB/ENC Training and Equipment

INTERVENTIONS:
Behavioral: HBB/ENC Training and Equipment — See the detailed description section
  Arms: Facilitators; Learners; Master Trainers
Other: HBB/ENC supplies — Staffs associated with participating facilities receive HBB/ENC training and use related equipment.
  Arms: Facilities

SUMMARY:
The primary purpose of this pre-post evaluation is to test the impact on perinatal mortality (fresh stillbirths or early neonatal deaths) among births > 1500g of training birth attendants at health facilities in the Helping Babies Breathe (HBB) and Essential Newborn Care (ENC) curricula. These facilities are located within clusters in the Global Network for Women's and Children's Health Research sites in Belgaum and Nagpur, India, and Eldoret, Kenya.

DETAILED DESCRIPTION:
Helping Babies Breathe (HBB) is a training program designed to resuscitate neonates regardless of where they were born. HBB was developed by the American Academy of Pediatrics (AAP), the NICHD's Global Network for Women's and Children's Health (GN), the Laerdal Foundation and their global partners. The HBB program was developed based upon the experience and results of an earlier Neonatal Resuscitation Program and the GN's FIRST BREATH randomized control trial.

The goal of the study is to test the impact of training birth attendants at selected health facilities in the Helping Babies Breathe (HBB) and Essential Newborn Care (ENC) curricula upon perinatal mortality (fresh stillbirths and early neonatal deaths), among births of ≥1500g. The training will take place in three GN sites, Kenya, and Nagpur and Belgaum, India. The study facilities serve the population in identified study clusters, defined geographic areas which participate in the GN's Maternal Newborn Health (MNH) Registry. In addition to measuring perinatal mortality rate pre and post training, the study will also assess resuscitation skills among the birth attendants as a result of the training. Quality Improvement activities are planned to ensure the integrity of the training, maintenance and availability of resuscitation equipment and skills maintenance.

The GN MNH Registry (NCT 01073475) was established in 2008 and includes all pregnancies and neonatal outcomes in defined geographic clusters. The primary outcome for the pre-post HBB evaluation study will be calculated using all delivery data from the GN MNH Registry for participating clusters during the defined study period.

The pre-post HBB evaluation will include the following key activities:

1. Selection of Master Trainers, Facilitators, and Learners
2. Country-level training of Master Trainers in the HBB and ENC curricula
3. Facility-level training of birth attendants in the HBB and ENC curricula
4. Periodic re-training of birth attendants in the HBB and ENC curricula
5. Quality improvement activities:

   * Regular observation of deliveries in participating study health facilities
   * Unannounced observation of deliveries (or HBB skills using a neonatal simulator if no deliveries are available)
   * Resuscitation debriefings
   * Perinatal Death audits
   * Daily bag and mask ventilation practice
   * Drills to practice emergency drills
   * Daily check of cleanliness and availability of resuscitation equipment.

The HBB Master Trainers (MT), Facilitators, and Learners will be evaluated at several points during the implementation of the training program and quality improvement activities.

ELIGIBILITY:
Inclusion Criteria:

* Facilities:

  * at least 60 deliveries per year;
  * ability to provide 24-hour coverage, 7 days per week in the delivery ward; and
  * minimum perinatal mortality rate of 30 per 1000 deliveries in the reference period.

Master Trainers (MT)

* Experienced teachers and content experts in neonatal resuscitation
* Trained and/or experienced in education
* Dedication to learner-focused education
* Able to give informed consent

Facilitators

* Experienced in teaching Learners in small groups
* Experienced in care of newborns
* Demonstrated understanding of course content
* Aptitude for teaching
* Able to give informed consent

Learners

* Skilled birth attendants with clearly defined responsibilities for attending deliveries at participating facilities
* Able to give informed consent

Exclusion Criteria:

* If a facility, master trainer, facilitator, or learner does not meet the above inclusion criteria they are excluded from the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70704 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Perinatal Mortality | Perinatal mortality data collected at 6 weeks post-delivery. Comparison will include the pre-intervention period of 12 months and the post-intervention period of 12 months.
  The difference in the rate of perinatal mortality (fresh stillbirth or neonatal death prior to 7 days) among births ≥1500g, pre versus post implementation of an integrated package of HBB and ENC training and equipment (referred to as HBB/ENC training and equipment). This measure will be calculated using delivery data from the Global Network's Maternal Newborn Health Registry for participating clusters.

SECONDARY OUTCOMES:
Facility-based perinatal mortality | Perinatal mortality data collected at 6 weeks post-delivery. Comparison will include the pre-intervention period of 12 months and the post-intervention period of 12 months.
  The difference in the rate of facility-based perinatal mortality, among births ≥1500g pre versus post implementation of HBB/ENC training and equipment.
Retention of resuscitation knowledge and skills | Assessments completed at initial training and refresher training.
  The difference pre versus post intervention in mean scores on a multiple choice test of resuscitation knowledge, observed skills in bag and mask ventilation (BMV), and OSCE A and OSCE B scenarios.
Number of neonatal resuscitations | Resuscitation data collected at 6 weeks post-delivery.
  The difference in the number of neonatal resuscitations, among births ≥1500g with bag and mask in participating facilities pre versus post HBB/ENC training and equipment.
Delivery room checklist score | Observations conducted on a monthly basis.
  The difference in scores on delivery room checklist (in facilities with > 100 deliveries/year)
Asphyxia related perinatal mortality | Perinatal mortality data collected at 6 weeks post-delivery. Comparison will include the pre-intervention period of 12 months and the post-intervention period of 12 months.
  The difference in the rate of asphyxia related perinatal mortality, among births ≥1500g pre versus post HBB/ENC training.
Health seeking behavior | Data collected at 6 weeks post-delivery. Comparison will include the pre-intervention period of 12 months and the post-intervention period of 12 months.
  The difference in the proportion of health seeking behavior pre versus post HBB/ENC training.
Facility deliveries | Data collected at 6 weeks post-delivery. Comparison will include the pre-intervention period of 12 months and the post-intervention period of 12 months.
  The difference in the proportion of facility deliveries pre versus post HBB/ENC training.
Very early newborn death (within 1 day of birth) | Data collected at 6 weeks post-delivery. Comparison will include the pre-intervention period of 12 months and the post-intervention period of 12 months.
  The difference in very early newborn death (within 1 day of birth) pre versus post HBB/ENC training.

CONTACTS AND LOCATIONS:
Overall Officials: Linda L. Wright, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (3):
- India (2):
  - Jawaharlal Nehru Medical College, Belagavi
  - Lata Medical Research Foundation, Nagpur
- Moi University School of Medicine, Eldoret, Kenya

REFERENCES:
- [Derived] Patel A, Bang A, Kurhe K, Bhargav S, Prakash A, Arramraj S, Hibberd PL. Comparison of perinatal outcomes in facilities before and after Global Network's Helping Babies Breathe Implementation Study in Nagpur, India. BMC Pregnancy Childbirth. 2019 Sep 4;19(1):324. doi: 10.1186/s12884-019-2480-7. PMID 31484498
- [Derived] Bang A, Patel A, Bellad R, Gisore P, Goudar SS, Esamai F, Liechty EA, Meleth S, Goco N, Niermeyer S, Keenan W, Kamath-Rayne BD, Little GA, Clarke SB, Flanagan VA, Bucher S, Jain M, Mujawar N, Jain V, Rukunga J, Mahantshetti N, Dhaded S, Bhandankar M, McClure EM, Carlo WA, Wright LL, Hibberd PL. Helping Babies Breathe (HBB) training: What happens to knowledge and skills over time? BMC Pregnancy Childbirth. 2016 Nov 22;16(1):364. doi: 10.1186/s12884-016-1141-3. PMID 27875999
- [Derived] Bellad RM, Bang A, Carlo WA, McClure EM, Meleth S, Goco N, Goudar SS, Derman RJ, Hibberd PL, Patel A, Esamai F, Bucher S, Gisore P, Wright LL; HBB Study Group. A pre-post study of a multi-country scale up of resuscitation training of facility birth attendants: does Helping Babies Breathe training save lives? BMC Pregnancy Childbirth. 2016 Aug 15;16(1):222. doi: 10.1186/s12884-016-0997-6. PMID 27527831
- [Derived] Bang A, Bellad R, Gisore P, Hibberd P, Patel A, Goudar S, Esamai F, Goco N, Meleth S, Derman RJ, Liechty EA, McClure E, Carlo WA, Wright LL. Implementation and evaluation of the Helping Babies Breathe curriculum in three resource limited settings: does Helping Babies Breathe save lives? A study protocol. BMC Pregnancy Childbirth. 2014 Mar 26;14:116. doi: 10.1186/1471-2393-14-116. PMID 24670013